CLINICAL TRIAL: NCT03352648
Title: CarDiac MagnEtic Resonance for Primary Prevention Implantable CardioVerter DebrillAtor ThErapy: an International Registry
Brief Title: CarDiac MagnEtic Resonance for Primary Prevention Implantable CardioVerter DebrillAtor ThErapy: an International Registry (DERIVATE)
Acronym: DERIVATE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Gianluca Pontone, MD, PhD (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Gianluca Pontone, MD, PhD, Director of MR Unit & Deputy Director of Cardiovascular CT Unit, Centro Cardiologico Monzino
Organization: Centro Cardiologico Monzino (Other)
Other Study IDs: R659/17-CCM698
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The DERIVATE study was conceived to integrate the information resulted from clinical data, transthoracic echocardiography, and cardiac magnetic resonance (CMR) imaging to provide a more reliable risk stratification in patients affected by heart failure (HF) and worthy of prophylactic implanted cardioverter defibrillator (ICD) therapy. The main purposes of this multicenter registry are to: 1) determine CMR findings, and specifically late gadolinium enhancement (LGE) features, T1 mapping, and extracellular volume (ECV) that predict sudden cardiac death (SCD) and ventricular arrhythmia; 2) provide a comprehensive clinical and imaging score that effectively improves the selection of patients who deserve a prophylactic ICD therapy; 3) evaluate the contribution of machine learning to predict major adverse cardiac events (MACE) as compared to standard clinical scores.

DETAILED DESCRIPTION:
The current guidelines provide indications for primary prevention implanted cardioverter defibrillator (ICD) therapy based on left ventricle ejection fraction (LVEF) and New York Heart Association (NYHA) class. This strategy is able to intercept only part of fatal arrhythmic events and, on the other hand, led to useless ICD implantations mainly among those patients with severe heart failure (HF) who will never incur in sever arrhythmias but rather will die because of decompensated HF. Cardiac magnetic resonance offers the possibility of identifying and quantitatively assessing myocardium fibrosis both localized in a specific area and diffuse and has already proved a significant prognostic meaning. DERIVATE is a prospective, international, multicenter, observational registry of stable HF patients with reduced LVEF who underwent clinical evaluation, transthoracic echocardiography (TTE) and cardiac magnetic resonance (CMR). Specifically, the primary aim of DERIVATE is to determine CMR findings that predict outcomes, with incremental value over LVEF and NYHA classification.

The DERIVATE registry uses a collaborative design with contribution and merger of similar prospectively enrolled cohorts from 33 sites in 6 countries in Europe and North America. The targeted population for the DERIVATE registry is a large sample of patients with clinical history of chronic HF who have undergone CMR by referral physician. Indication for CMR exams was recorded and classified according to the known causes of HF. All DERIVATE study patients are followed for all-cause mortality, sudden cardiac death (SCD), cardiovascular death (including death caused by acute myocardial infarction and stroke), sustained ventricular tachycardia (VT), aborted SCD, hospitalization or cardiac death related to chronic HF. The follow up minimum period is 12 months. Complete risk factors, clinical presentation, echocardiography and CMR data recording, and follow-up for all-outcomes will contribute data for common analysis.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure patients (according to the ACC/AHA classification) with known ischemic cardiomyopathy (ICM) or non ischemic dilated cardiomyopathy (DCM)
* reduced left ventricle ejection fraction (LVEF) (<50%)

Exclusion Criteria:

* pregnancy
* current alcohol or drug abuse
* unstable angina
* decompensated HF (NYHA class IV) in the previous 1 month
* acute myocarditis in the previous 3 months
* recent myocardial infarction (MI) (<40 days) or)
* severe valvular disease
* cardiac amyloidosis
* hypertrophic cardiomyopathy
* arrhthmogenic right ventricular cardiomyopathy
* takotsubo cardiomyopathy
* congenital heart disease
* non CMR compatible device
* estimated glomerular filtration rate ≤30 mL/min/1.73m2
* other contraindication to gadolinium contrast agent
* severe claustrophobia
* participating in other trials with an active treatment arm (not to exclude patients who are in trials of diagnostic techniques or approved therapies)
* unwilling or unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consist of patients at multiple international centers undergoing clinically-indicated cardiac magnetic resonance (CMR) as part of their standard of care.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | The follow up minimum period is 12 months

SECONDARY OUTCOMES:
sudden cardiac death (SCD) | The follow up minimum period is 12 months
aborted sudden cardiac death (SCD) | The follow up minimum period is 12 months
heart failure (HF) death | The follow up minimum period is 12 months
sustained ventricular tachycardia (VT) | The follow up minimum period is 12 months
major adverse cardiac events (MACE) | The follow up minimum period is 12 months
  composite end point of SCD, aborted SCD, cardiovascular death, and sustained VT

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Pontone, MD, Principal Investigator — IRCCS Centro Cardiologico Monzino, Milano, Italy; Andrea Igoren Guaricci, MD, Principal Investigator — University Hospital Policlinico Consorziale of Bari, Bari , Italy; Jurg Schwitter, MD, Principal Investigator — Lausanne University Hospital-CHUV, Lausanne, Vaud, Switzerland; Pier Giorgio Masci, MD, Principal Investigator — Lausanne University Hospital-CHUV, Lausanne, Vaud, Switzerland
Locations (29):
- United States (2):
  - Loyola University of Chicago,, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
- KU Leuven-University of Leuven, Leuven, Belgium
- St.Luke's Hospital Thessaloniki, Thessaloniki, Greece
- Italy (21):
  - Ospedale Medico-Chirurgico Accreditato Villa dei Fiori, Acerra
  - University Hospital Policlinico Consorziale, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - A.O. Desio e Vimercate - P.O. Desio, Desio
  - Ospedali Riuniti University Hospital, Foggia
  - University of Messina, Messina
  - IRCCS Policlinico San Donato,, Milan
  - Vita-Salute San Raffaele University, Milan
  - Centro Cardiologico Monzino, IRCCS, Milan
  - IRCCS Istituto Auxologico Italiano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - University of Padua, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Policlinico San Matteo Pavia Fondazione IRCCS, Pavia
  - Fondazione G. Monasterio CNR, Regione Toscana, Pisa
  - Azienda Unità Sanitaria Locale di Rimini - Regione Emilia Romagna, Rimini
  - Casilino Polyclinic, Roma
  - Vannini Hospital Rome, Roma
  - Sapienza University of Rome, Rome
  - Humanitas Research Hospital, Hospital Care and Research Institution, IRCCS,, Rozzano
  - University of Siena, Siena
- Lausanne University Hospital-CHUV, Lausanne, Switzerland
- United Kingdom (3):
  - Bristol Heart Institute, Bristol
  - King's College London, London
  - The Heart Hospital, London

REFERENCES:
- [Derived] Ghanbari F, Joyce T, Lorenzoni V, Guaricci AI, Pavon AG, Fusini L, Andreini D, Rabbat MG, Aquaro GD, Abete R, Bogaert J, Camastra G, Carigi S, Carrabba N, Casavecchia G, Censi S, Cicala G, De Cecco CN, De Lazzari M, Di Giovine G, Di Roma M, Focardi M, Gaibazzi N, Gismondi A, Gravina M, Lanzillo C, Lombardi M, Lozano-Torres J, Masi A, Moro C, Muscogiuri G, Nese A, Pradella S, Sbarbati S, Schoepf UJ, Valentini A, Crelier G, Masci PG, Pontone G, Kozerke S, Schwitter J. AI Cardiac MRI Scar Analysis Aids Prediction of Major Arrhythmic Events in the Multicenter DERIVATE Registry. Radiology. 2023 May;307(3):e222239. doi: 10.1148/radiol.222239. Epub 2023 Mar 21. PMID 36943075
- [Derived] Guaricci AI, Masci PG, Muscogiuri G, Guglielmo M, Baggiano A, Fusini L, Lorenzoni V, Martini C, Andreini D, Pavon AG, Aquaro GD, Barison A, Todiere G, Rabbat MG, Tat E, Raineri C, Valentini A, Varga-Szemes A, Schoepf UJ, De Cecco CN, Bogaert J, Dobrovie M, Symons R, Focardi M, Gismondi A, Lozano-Torres J, Rodriguez-Palomares JF, Lanzillo C, Di Roma M, Moro C, Di Giovine G, Margonato D, De Lazzari M, Perazzolo Marra M, Nese A, Casavecchia G, Gravina M, Marzo F, Carigi S, Pica S, Lombardi M, Censi S, Squeri A, Palumbo A, Gaibazzi N, Camastra G, Sbarbati S, Pedrotti P, Masi A, Carrabba N, Pradella S, Timpani M, Cicala G, Presicci C, Puglisi S, Sverzellati N, Santobuono VE, Pepi M, Schwitter J, Pontone G. CarDiac magnEtic Resonance for prophylactic Implantable-cardioVerter defibrillAtor ThErapy in Non-Ischaemic dilated CardioMyopathy: an international Registry. Europace. 2021 Jul 18;23(7):1072-1083. doi: 10.1093/europace/euaa401. PMID 33792661
- [Derived] Guaricci AI, Masci PG, Lorenzoni V, Schwitter J, Pontone G. CarDiac MagnEtic Resonance for Primary Prevention Implantable CardioVerter DebrillAtor ThErapy international registry: Design and rationale of the DERIVATE study. Int J Cardiol. 2018 Jun 15;261:223-227. doi: 10.1016/j.ijcard.2018.03.043. Epub 2018 Mar 11. PMID 29550015